CLINICAL TRIAL: NCT00528853
Title: Correlation of Lung Biopsy, BAL, and High Resolution CT Scan in Lung Transplantation. Can We Help Diagnose Acute Rejection and Better Predict Bronchiolitis Obliterans?
Brief Title: Correlation of Lung Biopsy, BAL, and High Resolution CT Scan in Lung Transplantation
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 15660A
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Bronchiolitis Obliterans Syndrome
Keywords: Bronchiolitis Obliterans Syndrome
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A major source of graft failure and dysfunction in lung transplantation is known to be bronchiolitis obliterans (BO)and its clinical correlate called bronchiolitis obliterans syndrome(BOS). In fact, BOS is the leading cause of death in lung recipients beyond one year post transplant. Currently, our ability to assess lung injury after transplant is less than ideal.

The purpose of this study is to use new computerized tomography(CT) technology, specifically , 64 bit acquisition, to detect and predict the onset of lung injuries, with the hope of finding better therapies that currently exist.

DETAILED DESCRIPTION:
Total enrollment : 10

Lung transplant patients will undergo CT Scans before scheduled bronchoscopies which are routinely performed at 1, 3, 6, 9, and 12 months post transplant. Imaging will be done with the newest generation scanner, with intent to analyze all pertinent areas of the lung for pathology, but especially the bronchial anastomoses, the lung parenchyma with focus on gas exchanging lobules of the lung, and any suspected abnormalities from physical exam, laboratory tests, or prior chest xray.

CT imaging will precede bronchoscopy and biopsy so that CT interpretation will be unencumbered by changes due to the bronchoscopic procedure.

ELIGIBILITY:
Inclusion Criteria:

* Lung transplant patients who are at least 18 years of age.
* All patients must be able to give written informed consent.

Exclusion Criteria:

* Lung transplant patients who are unable to undergo a CT Scan.
* Lung transplant patients who are unable to give informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung transplant patients meeting inclusion criteria will be recruited from the lung transplant clinic.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2007-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Garrity, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago Medical Center, Chicago, Illinois, United States